CLINICAL TRIAL: NCT03853629
Title: Reducing the Effects of Air Pollution on Children With Cystic Fibrosis
Brief Title: Air Pollution and Children With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 215879
Record Dates: First submitted 2019-02-19; First posted 2019-02-25 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2018-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CF: * Age 1-17
  * Diagnosis of Cystic Fibrosis
  * Living in or around London
  Interventions: Other: None. Not applicable
- Controls: * Age 1-17
  * Healthy
  * Living in or around London
  Interventions: Other: None. Not applicable

INTERVENTIONS:
Other: None. Not applicable — None. Not applicable

SUMMARY:
1. To determine personal exposure to air pollution in children with cystic fibrosis;
2. To determine airway macrophage uptake of inhaled particulate matter in cystic fibrosis children;
3. To establish whether prostaglandin E2 affects particulate matter removal in airway.

DETAILED DESCRIPTION:
Background:

Cystic fibrosis (CF) is the commonest hereditary life-shortening respiratory condition, resulting in premature death secondary to recurrent airway infections and inflammation, leading to irreversible lung damage. The screening programme in infancy has improved life expectancy but the lifespan of CF patients is still reduced by 20 years at present. Thus interventions to reduce inflammation, infection and lung damage in CF are still needed.

One potential intervention is to reduce exposure of CF children to air pollution. Particulate matter (PM) are microscopic soot particles from petrol and diesel engine emissions; PM is linked to adverse respiratory health effects in children. Children with cystic fibrosis are particularly vulnerable to PM but, to date, no exposure-reduction advice is available, and the mechanism underlying this vulnerability is unclear.

Personal exposure of CF children to PM is due to: i) locally-generated sources (relative to the proximity to busy roads) and ii) background concentrations (i.e. PM blown across the whole city from other areas). Although a link between air pollution and reduced lung function growth in healthy children is well established, the link with CF lung disease has only recently emerged. A recent study found that long-term exposure of CF children to PM increases risk of airway infection with Pseudomonas. Another study also found that short-term background pollution is associated with increased need for antibiotics in children and adults with CF. The need to reduce patients' personal exposure to PM has been recognised by Barts Health NHS Trust. Working with Global Action Plan, the Trust has developed tips on how to reduce adults' personal exposure to air pollution. These tips include traveling outside rush hours, taking low pollution routes (maps provided), and signing up to the airText air pollution warning App. Since travel outside rush hours is not feasible for school children, child-friendly tips are urgently needed.

Recent research in asthma patients suggests a putative mechanism of impaired removal of inhaled PM. In the healthy lung, inhaled PM is quickly removed (phagocytosed) by airway macrophages (AM). AM patrol the surface of epithelial cells lining the airways; after taking up PM, they move up and out of the lung. Thus AM with normal phagocytic function act to both reduce PM exposure of other airway cells - including epithelial cells, and to ensure that PM does not accumulate in the lung. The amount of carbon particles in AM was previously used to assess the effects of long-term effects of exposure of healthy children and adults. The amount of black carbon (BC) in AM reflects the intrinsic capacity of AM to remove PM (phagocytic capacity). AM carbon is significantly lower in conditions such as severe asthma, where AM phagocytic capacity is impaired. Furthermore, a role for prostaglandin E2 (PGE2) in mediating impaired phagocytic function in asthma has been identified. First, PGE2 suppresses AM phagocytosis of urban PM in vitro; and second, children with severe asthma had increased urinary PGE2 metabolites. Shift of inhaled PM away from AM to other cells has the potential to stimulate interleukin-8 (IL-8) release by epithelial cells - a phenomenon observed in mouse, where inhalation of non-inflammatory particles produces significant airway neutrophilia when AM phagocytic function is impaired.

The hypothesis is that impaired handling of inhaled PM by AM contributes to vulnerability of children with CF to air pollution. Specifically, increased vulnerability to inhaled PM in children with CF is due to PGE2-mediated impairment of AM phagocytosis. The corollary is that children with CF will have; i) reduced levels of AM carbon in vivo (reflecting reduced phagocytosis of inhaled PM in vivo), ii) reduced capacity of AM to phagocytose carbon PM in vitro, iii) increased metabolites of PGE2 in the airway and urine, and finally, iv) since PGE2 production is under the control of the enzyme cyclooxygenase (COX, especially COX-2), CF airway cells have increased COX-2 expression, v) COX inhibitors (e.g. Ibuprofen) should suppress PGE2 production, theoretically improving AM function.

Non-cystic fibrosis bronchiectasis is a respiratory condition with multiple aetiology such as congenital pathology, immunodeficiency, and primary ciliary dyskinesia. Patients with non-CF bronchiectasis demonstrate similar clinical features to those with CF, patients with either conditions are managed with similar treatments, it is therefore hypothesised that the above also apply to children with non-CF bronchiectasis.

There has been evidence that some organisms are capable of reproducing and residing within airway macrophages without being destroyed by the traditional phagocytic pathway. Often, unwell CF and non-CF bronchiectasis patients are admitted to the hospital for intensive antibiotic treatments but a proportion of their sputum samples yield no growth by routine hospital culture. This study will explore isolated airway macrophages and identify the organisms within - if any are present.

Clinical Data:

There is evidence to support this hypothesis; i) it was previously reported that phagocytosis of inert latex beads is impaired in AM from CF adults (71 + 15 % phagocytosis in controls vs. 23 + 9 % in CF), ii), CF is associated with increased airway PGE2, and iii) in a pilot study, significantly (p<0.01) reduced AM carbon in 6 CF children compared with 6 healthy controls (mean 0 vs. 0.3 + .05, μm2 p<0.01) was found.

Rationale:

To date, the effect of impaired uptake of PM by AM on other airway cells has not been studied in vitro. The hypothesis is that in co-cultures of human AM and airway epithelial cells exposed to urban PM, PGE2-mediated impairment of macrophage phagocytosis increases epithelial release of IL-8. Furthermore, since AM are a major source of airway PGE2, it is speculated that there is increased COX-2 expression in AM from CF children. Thus suppression of AM phagocytic function in CF is an autocrine process; i.e. CF AM release more PGE2 - which in turn suppresses AM phagocytosis. In this study the evidence will be sought for abnormal handling of PM by AM from CF children, and model this using cultures of human airway cells and macrophages.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-17
* Diagnosis of Cystic Fibrosis
* Diagnosis of non-CF bronchiectasis
* Living in or around London With age matched healthy controls

Exclusion Criteria:

* Current active smoker
* Receiving immunosuppressive drug therapy
* For children with CF not on regular nebulised hypertonic saline: drop in FEV1 of >15% post-bronchodilator (exclusion criterion for sputum induction)
* For healthy controls: Post-bronchodilator FEV1 <80% (standard exclusion criterion for sputum induction in healthy individuals)
* For participants currently or recently involved in other research study, they will be excluded if their current or recent research have any potential impact on our sampling or results.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Inclusion Criteria:
  * Age 1-17
  * Diagnosis of Cystic Fibrosis
  * Diagnosis of non-CF bronchiectasis
  * Living in or around London With age matched healthy controls
  Exclusion Criteria:
  * Current active smoker
  * Receiving immunosuppressive drug therapy
  * For children with CF not on regular nebulised hypertonic saline: drop in FEV1 of >15% post-bronchodilator (exclusion criterion for sputum induction)
  * For healthy controls: Post-bronchodilator FEV1 <80% (standard exclusion criterion for sputum induction in healthy individuals)
  * For participants currently or recently involved in other research study, they will be excluded if their current or recent research have any potential impact on our sampling or results.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Airway macrophage uptake of inhaled particulate matter in both groups of children | 3 years
  Black carbon loading area (micro-square meters) of airway macrophages, using light microscopy

SECONDARY OUTCOMES:
Personal exposure to air pollution in both groups of children | 3 years
  Black carbon level (nanograms per cubic meter) of children's personal exposure - using an aethalometer.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Grigg, Principal Investigator — Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No